CLINICAL TRIAL: NCT00969943
Title: Gender Differences in Response to Cues in Cocaine Dependence
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Kathleen Brady, MD, PhD, Distinguished University Professor, Medical University of South Carolina
Other Study IDs: 10598
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Cocaine Dependence
Keywords: HPA axis
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Cocaine-dependent Men
- Cocaine-dependent Women
- Control Men
- Control Women

SUMMARY:
The purpose of this study is to evaluate whether men and women respond differently to seeing items related to cocaine use or to remembering stressful events. Four groups of individuals will be recruited to participate in this study: men with cocaine dependence, women with cocaine dependence, men without cocaine dependence, and women without cocaine dependence.

Hypothesis #1: Cocaine-dependent women will demonstrate smaller increases in neuroendocrine, but greater increases in heart rate and more cocaine craving and subjective distress when exposed to stress as compared to cocaine-dependent men and non cocaine-dependent men and women.

Hypothesis #2: Cocaine-dependent men will demonstrate greater increases in neuroendocrine, but greater increases in heart rate and more cocaine craving and subjective distress when exposed to cocaine-related cues as compared to cocaine-dependent women and non cocaine-dependent men and women.

Hypothesis #3: Cocaine-dependent women will demonstrate greater increases in heart rate and more cocaine craving and subjective distress when exposed to stress inducing stimuli as compared to their own responses to a cocaine-related cue.

Hypothesis #4: The neuroendocrine response to a stress hormone (corticotropin releasing hormone; CRH) will be greater in cocaine-dependent women as compared to cocaine-dependent men.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
* Subjects must consent to remain abstinent from all drugs of abuse (except nicotine) for a two-day period immediately prior to the GCRC admission. In cases where lab results, subject self-report, or staff observation suggests that a patient has used alcohol or drugs within two days of hospital admission, the patient will be admitted at the discretion of on-call study staff. Nicotine dependence can affect HPA function (Baron et al., 1995) therefore it would be ideal to exclude subjects with nicotine use from all four groups. Because of the high comorbidity of alcohol use and cocaine dependence, individuals with alcohol abuse or dependence will be included. Approximately equal numbers of nicotine-dependent individuals will be recruited into each of the study groups. Alcohol use for two days prior to testing will be discouraged, and nicotine use immediately prior to the testing session will be controlled.
* Subjects must consent to random assignment.
* Subjects must consent to outpatient admission at the GCRC and two overnight admissions at the Medical University Hospital.
* Subjects must consent to a one-week and one-month follow-up visit after the GCRC admission.

Exclusion Criteria:

* Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control. Because oral contraceptives may affect HPA axis function, the number of women on various types of oral contraceptives (triphasic vs static) and women on depot progesterone will be balanced between groups
* Women with premenstrual dysphoric disorder as this may impact on the response to the stress test procedure (Woods et al., 1994).
* Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease including diabetes, as these conditions may affect HPA axis function.
* Subjects with any liver function test (LFTs) of greater than two times normal, as compromised liver function can interfere with HPA axis activity (Williams & Dluhy, 1987).
* Subjects with Addison's disease, Cushing's disease or other diseases of the adrenal cortex likely to affect HPA axis function.
* Subjects with a history of or current psychotic disorder or bipolar affective disorder as these may interfere with HPA function.
* Subjects with current major depressive disorder or post-traumatic stress disorder as these disorders are associated with characteristic changes in HPA axis function.
* Subjects receiving synthetic glucocorticoid therapy, any exogenous steroid therapy, or treatment with other agents that interfere with HPA axis function within one month of the time of testing.
* Subjects taking opiates, opiate antagonists, or benzodiazepines. (Subjects who have been maintained on SSRI's, anticonvulsants, or antipsychotics (for sleep only) for more than 8 weeks or longer are NOT excluded).
* Subjects with any acute illness or fever as this may affect HPA axis activity. Individuals who otherwise meet study criteria will be rescheduled for evaluation for participation.
* Subjects who are 30% over ideal weight or have a BMI greater than 30 will be considered for study participation based on the clinical judgment of study staff.
* Subjects who are unwilling to maintain abstinence from alcohol and other drugs of abuse (except nicotine) for two days prior to the stress task procedure.
* Women who gave birth to a child within the past 6 months of initial screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be four primary sources of recruitment for cocaine dependent subjects: (1) patients referred from the Center for Drug and Alcohol Programs (CDAP) intake coordinator, (2) individuals presenting to CDAP for either inpatient or outpatient treatment, (3) individuals presenting to the Charleston Center for inpatient or outpatient treatment, (4) and individuals presenting to the Dorchester Alcohol and Drug Commission (DADC) for treatment. Control subjects will be recruited from the Charleston community
Sampling Method: Non-Probability Sample
Dates: Start 2003-03 (Actual); Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- MUSC-Clinical Neurosciences Division, Charleston, South Carolina, United States

REFERENCES:
- [Result] Brady KT, McRae AL, Moran-Santa Maria MM, DeSantis SM, Simpson AN, Waldrop AE, Back SE, Kreek MJ. Response to corticotropin-releasing hormone infusion in cocaine-dependent individuals. Arch Gen Psychiatry. 2009 Apr;66(4):422-30. doi: 10.1001/archgenpsychiatry.2009.9. PMID 19349312